CLINICAL TRIAL: NCT04771559
Title: Evaluation of the Effect and Side Effect Profile of Covid-19 Vaccine in Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Ayşe İrem Yasin, MD, Bezmialem Vakif University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 132620
Record Dates: First submitted 2021-02-17; First posted 2021-02-25 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Covid19; Cancer
Keywords: Cancer, Covid-19, Vaccine
MeSH Terms: conditions — COVID-19; Neoplasms | interventions — COVID-19 Serological Testing

STUDY DESIGN:
Intervention Model Description: The study consists of two groups : 1) Cancer patients, 2) Healthy controls Blood samples will be taken from the participants of the two groups 4 weeks after the second dose of the COVID-19 vaccine and antibody testing will be performed. Additionally participants will be questioned for side effects of the vaccine and the data will be registered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cancer patients (Other): Covid-19 antibody levels of patients will be measured
  Interventions: Other: COVID-19 antibody test
- Healthy control (Other): Covid-19 antibody levels of healthy controls will be measured
  Interventions: Other: COVID-19 antibody test

INTERVENTIONS:
Other: COVID-19 antibody test — 5 cc blood sample from each participant will be taken 4 weeks after the second dose of the COVID-19 vaccine . After blood samples are centrifuged at 2500 rpm for 10 minutes, the separated serum will be backed up in two different ependorphs and stored at -80 or -20 degrees. The samples will be delivered to the working center in a manner suitable for cold chain transport. COVID-19 antibody test will be performed on the blood samples

SUMMARY:
The aim of the study is to evaluate the effects and side effects of inactive COVID-19 vaccine in patients with cancer and compare them with the healthy control group.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the effects and side effects of inactive COVID-19 vaccine in patients with cancer. Patients followed up in medical oncology clinic and healthy volunteers will be enrolled in the study. Blood samples of participants will be taken 4 weeks after the second dose of the COVID-19 vaccine. After blood samples are centrifuged at 2500 rpm for 10 minutes, the separated serum will be backed up in two different eppendorf tubes and stored at -80 or -20 degrees. The samples will be delivered to the working center in a manner suitable for cold chain transport. COVID-19 antibody test will be performed on the blood samples. In addition, volunteers will be questioned in terms of side effects that may develop after vaccination and the information obtained will be recorded in the database together with the clinical data of the patients.

ELIGIBILITY:
Inclusion Criteria:

For the patient group :

1. Patients with pathological and clinical cancer diagnosis
2. Older than 18 years
3. Patients two doses of COVID-19 vaccine administered
4. Volunteering to participate in the study

For the control group :

1. No known cancer diagnosis or history
2. Older than 18 years
3. Two doses of COVID-19 vaccine administered
4. Volunteering to participate in the study -

Exclusion Criteria:

1. Not volunteering to participate in the study
2. < 18 years
3. Not administered two doses of the COVID-19 vaccine
4. Covid-19 infection history -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1500 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Antibody levels | 1 month
  COVID-19 antibody titers of the patients will be measured in blood samples.

SECONDARY OUTCOMES:
Side effects | 1 month
  Participants will be questioned for common side effects

CONTACTS AND LOCATIONS:
Overall Officials: MAHMUT GUMUS, PROF, Study Chair — MEDENIYET UNIVERSITY; AHMET BILICI, PROF, Study Chair — Medipol University; HACI MEHMET TURK, PROF, Study Chair — BEZMIALEM UNIVERSITY; MESUT SEKER, PROF, Study Director — BEZMIALEM UNIVERSITY; AYSE IREM YASIN, MD, Principal Investigator — BEZMIALEM UNIVERSITY; BILGE SUMBUL, ASOC.PROF., Study Chair — BEZMIALEM UNIVERSITY; FAYSAL DANE, PROF, Study Chair — Acibadem University; CAGLAYAN GEREDELI, ASOC.PROF., Study Chair — OKMEYDANI RESEARCH HOSPITAL
Locations (5):
- Turkey (Türkiye) (5):
  - Bezmialem University, Istanbul, Fatih
  - Okmeydani Research Hospital, Istanbul, Fatih
  - Acibadem University, Istanbul
  - Medeniyet University, Istanbul
  - Medipol University, Istanbul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yasin AI, Aydin SG, Sumbul B, Koral L, Simsek M, Geredeli C, Ozturk A, Perkin P, Demirtas D, Erdemoglu E, Hacibekiroglu I, Cakir E, Tanrikulu E, Coban E, Ozcelik M, Celik S, Teker F, Aksoy A, Firat ST, Tekin O, Kalkan Z, Turken O, Oven BB, Dane F, Bilici A, Isikdogan A, Seker M, Turk HM, Gumus M. Efficacy and safety profile of COVID-19 vaccine in cancer patients: a prospective, multicenter cohort study. Future Oncol. 2022 Mar;18(10):1235-1244. doi: 10.2217/fon-2021-1248. Epub 2022 Jan 27. PMID 35081732